CLINICAL TRIAL: NCT04267484
Title: Technology to Support Decision Making About Aging at Home (COORDINATEs)
Brief Title: What Are my Options to Stay Safe at Home: Technology For Aging at Home
Acronym: COORDINATEs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Dalarna University (Other); University of Groningen (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, France Legare, Principal investigator, CHU de Quebec-Universite Laval
Other Study IDs: 118792
Record Dates: First submitted 2020-02-07; First posted 2020-02-13 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Memory Problems; Aging; Mild Cognitive Impairment; Shared Decision Making
Keywords: Shared decision making; Mild Cognitive Impairment; Technology; aging in place; memory problem
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults with mild cognitive impairment: WP1, older adults with cognitive impairment will use a GPS tracker for 2 weeks, during which they are asked 1) to keep a daily diary about their activity (travel diary), 2) take the researcher on a walk that they often do (walking interview), and 3) participate in an in-depth interview after 2 weeks, in which their experience with the GPS ans the travel diary data are discussed.
  WP2, older adults with mild cognitive impairment, caregivers, health professionals and technology developers will collaborate during group discussion meeting to co-design the e-decision support platform to be adapted.
  WP3, older adults with mild cognitive impairment, caregivers and health professionals will then be asked to use the adapted e-decision support platform and fill a survey.
  Interventions: Device: GPS and travel diary; Other: e-decision support platform

INTERVENTIONS:
Device: GPS and travel diary — WP1: GPS tracker for 2 weeks and a daily diary about activity (travel diary).
Other: e-decision support platform — WP2 and WP3: An e-decision support platform that will foster shared decision making about options to stay safe at home for the older adult.

SUMMARY:
Most older people want to stay at home as long as possible. Effective self-management for people losing autonomy depends on reliable monitoring of their mobility, health and safety and active implication in decision-making. New technologies have the potential to provide information about changing patterns that reflect changing care needs. This information could help older adults, caregivers and health professionals to participate in decision-making about housing options when a change in living environment needs to be considered.

DETAILED DESCRIPTION:
This is a multi-phase study to be conducted in 3 countries: Canada (Quebec and Alberta), Sweden and Netherlands. The primary objective is to provide e-decision support technology that will facilitate self-management in the context of aging in place and foster informed value congruent decisions about options to age safely at home.

The aim of the project is to develop and validate a e-technology based on already existing components (e.g. GPS devices, diverse e-platforms and decision support interventions) to 1) help older adults with mild cognitive impairment/memory problems to stay safely at home as long as possible and 2) to provide older adults with decision support tools to help them make informed value congruent decisions (e.g. foster a shared decision-making process) regarding aging at home in a safe manner.

The secondary objectives are:

1. Assess autonomy and mobility of older adults with mild cognitive impairment/memory problems living at home.
2. Inform shared decision-making processes about options to safely age in place for all those involved.

The investigators will apply an integrated Knowledge Translation (iKT), comparative, mixed-methods approach to explore, older adults living at home with mild cognitive impairment/memory problems, their use of space in their homes and neighbourhoods.

The project is divide into 4 work package (WP). In more details, during WP1, the investigators will collect spatial data (e.g. using GPS) and self-reported data (e.g. travel diaries, walking interviews, in-depth interviews, surveys). At WP2, the investigators will use iterative end-user feedback and end-user consultation discussion group to tailor a decision support technology to knowledge-users. At WP3, investigators will assess user opinion regarding factors that could influence their use of the newly adapted e-decision support technology. Finally, at WP4 the investigators will triangulate data and take into account differences between jurisdictions.

This collaboration and our cross-country comparisons will contribute to scaling up e-decision support solutions in the future for the older adults with mild cognitive impairment/memory problems who want to age safely at home.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years
* Living at home
* Diagnosed with mild cognitive impairment or experiencing memory issues
* Able to read, understand and write
* Can provide informed consent

Exclusion Criteria:

* Older adults who are not able to provide informed consent
* Living in nursing home or hospital

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (>65 years) with mild cognitive impairment or self reported memory problems.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Autonomy and mobility assessment using GPS | Participant will wear a GPS for a total of two weeks. As data collection will occur in parallel at all four sites (Quebec, Alberta, Sweden, Netherlands) data collection will happen over a period of 1 year
  WP1: 1) Asses autonomy and mobility of older adults with mild cognitive impairment and memory problems living at home (including caregivers), their movement through their homes and neighborhoods (using GPS and walking interview); 2) how GPS data can support ongoing SDM about housing options for older adults.
Iterative assessment to tailor the e-decision support technology | Immediately after group discussion. 3 sequential group discussion are plan to occur, one in each country (Canada, Sweden, Netherlands) data collection will happen over a period of 1 year.
  WP2: 1) Group discussion on if and how to incorporate GPS and adaptation of an existing e-platforms to create an adapted e-decision support technology (noted that the discussion focus will depend on result from WP1).
User experience assessment of the newly adapted technology | Immediately after testing the new platform. As data collection will occur in parallel at all four sites (Quebec, Alberta, Sweden, Netherlands), it will happen over a period of 6 months
  WP3: 1) Opinion of older adults with mild cognitive impairment, caregivers and health professionals about the adapted technology (noted that the final survey will depend on result from WP1 and WP2).

SECONDARY OUTCOMES:
Inform SDM processes about housing option | 9 months
  WP4: 1) Knowledge about differences and similarities between three countries
Open-ended questionnaire of participant global health status and their experience of using the GPS and filling the travel diary | Immediately before and after carrying the GPS at WP1. As data collection will occur in parallel at all four sites (Quebec, Alberta, Sweden, Netherlands) data collection will happen over a period of 1 year
  WP1: Participant will be ask to share their experience with the GPS and the travel diary

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, PhD, Principal Investigator — Laval University
Locations (4):
- Canada (2):
  - CERSSPL, Québec, Quebec
  - University of Alberta, Edmonton
- University of Groningen, Groningen, Netherlands
- Dalarna University, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Caron CD, Ducharme F, Griffith J. Deciding on institutionalization for a relative with dementia: the most difficult decision for caregivers. Can J Aging. 2006 Summer;25(2):193-205. doi: 10.1353/cja.2006.0033. PMID 16821201
- [Result] Garvelink MM, Emond J, Menear M, Briere N, Freitas A, Boland L, Perez MMB, Blair L, Stacey D, Legare F. Development of a decision guide to support the elderly in decision making about location of care: an iterative, user-centered design. Res Involv Engagem. 2016 Jul 19;2:26. doi: 10.1186/s40900-016-0040-0. eCollection 2016. PMID 29062524
- [Result] Pot AM, Willemse BM, Horjus S. A pilot study on the use of tracking technology: feasibility, acceptability, and benefits for people in early stages of dementia and their informal caregivers. Aging Ment Health. 2012;16(1):127-34. doi: 10.1080/13607863.2011.596810. Epub 2011 Jul 25. PMID 21780960
- [Result] Greenhalgh T, Jackson C, Shaw S, Janamian T. Achieving Research Impact Through Co-creation in Community-Based Health Services: Literature Review and Case Study. Milbank Q. 2016 Jun;94(2):392-429. doi: 10.1111/1468-0009.12197. PMID 27265562
- [Result] Meijering L, Weitkamp G. Numbers and narratives: Developing a mixed-methods approach to understand mobility in later life. Soc Sci Med. 2016 Nov;168:200-206. doi: 10.1016/j.socscimed.2016.06.007. Epub 2016 Jun 8. PMID 27316320
- [Derived] Sturge J, Meijering L, Jones CA, Garvelink M, Caron D, Nordin S, Elf M, Legare F. Technology to Improve Autonomy and Inform Housing Decisions for Older Adults With Memory Problems Who Live at Home in Canada, Sweden, and the Netherlands: Protocol for a Multipronged Mixed Methods Study. JMIR Res Protoc. 2021 Jan 21;10(1):e19244. doi: 10.2196/19244. PMID 33475512
- See also: Chaire de recherche du Canada sur la décision partagée et l'application des connaissances — http://www.decision.chaire.fmed.ulaval.ca/